CLINICAL TRIAL: NCT02147249
Title: Inflammatory Proteins, Gene Polymorphisms, and Transcriptome Profiles in Patients With Erythema Migrans
Brief Title: Cytokines and Chemokines in Erythema Migrans
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Medical Centre Ljubljana (Other)
Collaborators: University of Ljubljana School of Medicine, Slovenia (Other); Medical University of Vienna (Other); Harvard University (Other)
Responsible Party: Principal Investigator, Franc Strle, MD, PhD, University Medical Centre Ljubljana
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: EM-0613
Record Dates: First submitted 2013-06-24; First posted 2014-05-26 (Estimated); Last update posted 2019-04-22 (Actual); Status verified 2019-04

CONDITIONS: Erythema Migrans
Keywords: erythema migrans; Lyme borreliosis; inflammation; outcome
MeSH Terms: conditions — Glossitis, Benign Migratory; Lyme Disease; Inflammation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- erythema migrans patients treated with antibiotics (Experimental): adult patients with erythema migrans will be treated with oral antibiotics
  Interventions: Drug: antibiotic treatment

INTERVENTIONS:
Drug: antibiotic treatment — Patient will be treated with: doxycycline orally, 100 mg, bid, 14 days or cefuroxime axetil orally, 500 mg, bid, 14 days or amoxicillin orally, 500 mg, tid, 14 days

SUMMARY:
The main objective of this study is to characterize the inflammatory proteins, gene polymorphisms, and transcriptome profiles in patients with erythema migrans to gain better insight into pathogenesis of early Lyme borreliosis and to define new immune modulators that could serve as biomarkers of disease activity.

ELIGIBILITY:
Inclusion Criteria:

* erythema migrans in patients > 18 years

Exclusion Criteria:

* pregnancy or lactation
* taking antibiotic with antiborrelial activity within 10 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2013-07; Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
inflammatory proteins in erythema migrans patients | up to 12 months follow-up
  The inflammatory immune profiles will be assessed using Luminex to measure the expression of cytokines and chemokines representative of innate and adaptive TH1, TH2, TH17, and B cell responses in serum and if available, skin, of patients during active infection and after treatment.

SECONDARY OUTCOMES:
gene polymorphisms in erythema migrans patients | at enrollment
  The expression of disease-relevant genomic variants will be assessed using ImmunoChip.

OTHER OUTCOMES:
transcriptome profiles in erythema migrans patients | at 6 month follow-up
  We will use RNA sequencing of individual immune cell subtypes from patients to determine their transcriptome.

CONTACTS AND LOCATIONS:
Overall Officials: Franc Strle, MD, PhD, Study Chair — UMC Ljubljana; Dasa Stupica, MD, PhD, Principal Investigator — UMC Ljubljana
Locations (1):
- UMC Ljubljana, Department of Infectious Diseases, Ljubljana, Slovenia